CLINICAL TRIAL: NCT04634500
Title: Therapeutic Confirmatory Study to Evaluate the Efficacy and Safety of DWP16001 in Combination With Metformin in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Metformin Alone
Brief Title: The Efficacy and Safety of DWP16001 in Combination With Metformin in Patients With Type 2 Diabetes.
Acronym: ENHANCE-M
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWP16001302
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: T2DM (Type 2 Diabetes Mellitus)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Enavogliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): DWP16001 A mg, Dapagliflozin placebo
  Interventions: Drug: Dapagliflozin
- Control group (Active Comparator): DWP16001 A mg placebo, Dapagliflozin
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin Tablet
  Other Names: DWP16001

SUMMARY:
Therapeutic Confirmatory Study to Evaluate the Efficacy and Safety of DWP16001 in Combination with Metformin in Patients With Type 2 Diabetes Mellitus who Have Inadequate Glycemic Control on Metformin Alone.

DETAILED DESCRIPTION:
A Multi-center, Randomized, Double-Blind, Active-controlled, Phase 3, Therapeutic Confirmatory Study to Evaluate the Efficacy and Safety of DWP16001 in Combination with Metformin in Patients With Type 2 Diabetes Mellitus who Have Inadequate Glycemic Control on Metformin Alone.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with T2DM aged 19 to 80 years
2. Subjects who have received metformin alone at a fixed dose for the last 8 weeks and has 7% ≤ HbA1c ≤ 10.5%
3. Subjects with BMI of 20-45 kg/m2
4. Subjects who voluntarily decided to participate and provided written consent after being told of the objectives, method, and effects of this study

Exclusion Criteria:

1. Subjects with current or history of hypersensitivity to the IP of this study, metformin or drugs of the same class and their components (e.g., history of hypersensitivity to biguanide or SGLT2 inhibitors)
2. Diabetic ketoacidosis, diabetic coma or precoma within the past year
3. Urinary tract infections or genital infections within
4. Uncontrolled hypertension (SBP > 180 mmHg or DBP > 110 mmHg)
5. eGFR < 60 mL/min/1.73 m2
6. Severe heart failure (NYHA class III/IV)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | at 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Daewoong pharmatceutical, Soeul, South Korea

REFERENCES:
- [Derived] Han KA, Kim YH, Kim DM, Lee BW, Chon S, Sohn TS, Jeong IK, Hong EG, Son JW, Nah JJ, Song HR, Cho SI, Cho SA, Yoon KH. Efficacy and Safety of Enavogliflozin versus Dapagliflozin as Add-on to Metformin in Patients with Type 2 Diabetes Mellitus: A 24-Week, Double-Blind, Randomized Trial. Diabetes Metab J. 2023 Nov;47(6):796-807. doi: 10.4093/dmj.2022.0315. Epub 2023 Feb 9. PMID 36756676